CLINICAL TRIAL: NCT02690974
Title: Prospective, Multi-center, Open lAbel, Post-appRovAl Study AImed at Characterizing the Use of LCZ696 at 97 mg Sacubitril / 103 mg Valsartan Bid in Patients With HFrEF
Brief Title: Description of Tolerability of LCZ696 (Sacubitril / Valsartan) in Heart Failure With Reduced Ejection Fraction (HFrEF) Treated in Real Life Setting
Acronym: PARASAIL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CLCZ696BCA02
Record Dates: First submitted 2016-02-15; First posted 2016-02-24 (Estimated); Results first posted 2019-06-07 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-03

CONDITIONS: Hearth Failure With Reduced Ejection Fraction (HFrEF)
Keywords: HFrEF,; ACEi,; ACE inhibitor,; ARBs,; systolic heart failure,; chronic heart failure,; CHF,; reduced EF,; Ejection Fraction
MeSH Terms: conditions — Heart Failure, Systolic | interventions — sacubitril and valsartan sodium hydrate drug combination; sacubitril; Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LCZ696 (sacubitril / valsartan) (Other): All patients were initiated on either LCZ696 at 24 mg sacubitril / 26 mg valsartan or LCZ696 at 49 mg sacubitril / 51 mg valsartan bid for 2-4 weeks and were up-titrated to the next higher dose for another 2 - 4 weeks as applicable.
  Interventions: Drug: LCZ696 (sacubitril/valsartan)

INTERVENTIONS:
Drug: LCZ696 (sacubitril/valsartan) — All patients were treated with the LCZ696 (sacubitril and valsartan) tablets

SUMMARY:
The primary purpose of the study was to describe the tolerability of treatment with the optimal dose of LCZ696 (97 mg sacubitril / 103 mg valsartan bid), over six (6) months, in patients with heart failure with reduced ejection fraction (HFrEF) in Canada.

The study was also to describe the overall tolerability, effectiveness and safety of LCZ696 for the management of HFrEF over 12 months of treatment, as well as describe the patterns of LCZ696 up and down dose titrations occurring during the management of patients with HFrEF.

ELIGIBILITY:
Key Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Age ≥ 18 years and ≤ 80 years.
3. Males or females.
4. Diagnosis of Heart Failure NYHA class II-III.
5. Diagnosis of Heart Failure with reduced Ejection Fraction (LVEF =< 40%) and NYHA class II or III.
6. Stable on any dose of ACEI or ARB prior to enrolment in the study
7. Stable on any dose of a beta-blocker prior to enrolment in the study.
8. Eligible for treatment with LCZ696 as per Canadian product monograph.
9. Treated as an outpatient.
10. Signed an informed consent agreeing to participate in the study.

Key Exclusion Criteria:

1. Symptomatic hypotension and/or a SBP < 100 mmHg at baseline visit.
2. Estimated GFR < 30 mL/min/1.73m^2 as measured by the simplified Modification of Diet in Renal Disease (MDRD) formula at baseline visit.
3. Known history of angioedema related to previous ACEI or ARBs therapy, or history of hereditary or idiopathic angioedema.
4. Requirement of concomitant treatment with both ACEIs and ARBs.
5. Concurrent participation in other clinical trials or receiving other investigational drugs within 30 days of enrollment.
6. Hypersensitivity to the active substances, sacubitril or valsartan, or to any of the excipients.
7. Concomitant use of aliskiren-containing drugs in patients with diabetes mellitus (type 1 or type 2) or moderate to severe renal impairment (GFR <60ml/min/1.73m^2).
8. History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes.
9. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
10. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
11. Women of childbearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception during dosing of study treatment. Effective contraception methods are described in the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2017-06-07 (Actual); Study Completion 2017-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (28):
- Canada (28):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, New Westminster, British Columbia
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, Moncton, New Brunswick
  - Novartis Investigative Site, St. John's, Newfoundland and Labrador
  - Novartis Investigative Site, Burlington, Ontario
  - Novartis Investigative Site, Cambridge, Ontario
  - Novartis Investigative Site, Greater Sudbury, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Mississauga, Ontario
  - Novartis Investigative Site, Newmarket, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Peterborough, Ontario
  - Novartis Investigative Site, Sarnia, Ontario
  - Novartis Investigative Site, Scarborough Village, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Waterloo, Ontario
  - Novartis Investigative Site, Weston, Ontario
  - Novartis Investigative Site, Greenfield Park, Quebec
  - Novartis Investigative Site, Joliette, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Saint-Jean-sur-Richelieu, Quebec
  - Novartis Investigative Site, Terrebonne, Quebec
  - Novartis Investigative Site, Brossard
  - Novartis Investigative Site, Hamilton
  - Novartis Investigative Site, Québec
  - Novartis Investigative Site, Saint-Lambert

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 32 study centers in Canada
Pre-assignment Details: Approximately 300 patients with HFrEF were planned for enrolling into the study. A total of 302 patients received at least one dose of LCZ696 and were included in the Full Analysis Set (FAS). The analysis of the primary endpoint was based on the FAS.
Period: Overall Study
Arm/Group | LCZ696 (Sacubitril / Valsartan)
Started (All enrolled patients to whom treatment had been assigned (FAS)) | 302
Completed | 262
Not Completed | 40
Not completed — Adverse Event | 16
Not completed — Death | 9
Not completed — Subject/guardian decision | 4
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal of Informed Consent | 3
Not completed — Physician Decision | 2
Not completed — Non-compliance with study treatment | 1
Not completed — Protocol-defined stopping criteria | 1
Not completed — Protocol Deviation | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS)
Arm/Group | LCZ696 (Sacubitril / Valsartan)
Number analyzed (Participants) | 302
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.47 (10.7659)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 240
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 271
  Black | 8
  Asian | 15
  Native American | 4
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants on LCZ696 200 mg Bid at Month 6
Description: The tolerability of LCZ696 was defined as the percentage of patients on LCZ696 at the dose of 97 mg sacubitril / 103 mg valsartan twice daily (bid) who did not experience down titration or treatment discontinuation because of adverse events while on this dose at month 6. Only descriptive analysis done.
Time Frame: Month 6
Population: The Full Analysis Set (FAS), which consisted of all participants with an observed value, was considered.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | LCZ696 (Sacubitril / Valsartan)
Number analyzed (Participants) | 302
Percentage of Participants | 64.6 [59.18 to 69.96]

2. Secondary Outcome: Percentage of Participants on LCZ696 200 mg Bid at Month 12
Description: The tolerability of LCZ696 was defined as the percentage of patients on LCZ696 at the dose of 97 mg sacubitril / 103 mg valsartan twice daily (bid) who did not experience down titration or treatment discontinuation because of adverse events while on this dose at month 12. Only descriptive analysis done.
Time Frame: Month 12
Population: The Full Analysis Set (FAS), which consisted of all participants with an observed value, was considered.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | LCZ696 (Sacubitril / Valsartan)
Number analyzed (Participants) | 302
Percentage of Participants | 62.3 [56.78 to 67.72]

3. Secondary Outcome: Percentage of Participants Requiring Down-titration From LCZ696 200 mg
Description: The impact of the titration scheme on the tolerability of patients maintained on LCZ696 97 mg sacubitril / 103 mg valsartan bid was defined as the percentage of patients on LCZ696 200mg requiring down-titration. Only descriptive analysis done.
Time Frame: Month 12
Population: The Full Analysis Set (FAS), which consisted of all participants with an observed value, was considered.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | LCZ696 (Sacubitril / Valsartan)
Number analyzed (Participants) | 302
Percentage of Participants | 11.92 [8.27 to 15.58]

4. Secondary Outcome: Percentage of Participants With Down-titration Changes From LCZ696 200 mg During 12 Months of Treatment
Description: The impact of the titration scheme on the tolerability of patients maintained on LCZ696 97 mg sacubitril / 103 mg valsartan bid was defined as the number of down-titration during the 12 months treatment period. Dow-titration schemes considered for the analysis are 200 mg to 100 mg; 100 mg to 50 mg; and 50 mg to 0 mg (i.e. treatment discontinuation). The down-titration scheme of 50mg to 0 mg was taken in account in this analysis to ensure to reflect all actual changes in dose. Only descriptive analysis done.
Time Frame: Month 12
Population: The Full Analysis Set (FAS), which consisted of all participants with an observed value, was considered.
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 (Sacubitril / Valsartan)
Number analyzed (Participants) | 302
Participants
  200 mg dose level | 188
  100 mg dose level | 44
  50 mg dose level | 28

5. Secondary Outcome: Change From Baseline in the Six Minute Walk Test (6MWT) at Month 6 and Month 12
Description: The impact of LCZ696 on functional exercise capacity was measured by the Six Minute Walk Test at 6 and 12 months. The 6MWT measures the distance an individual is able to walf over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is able to self-pace and rest as needed as they traverse back and forth along a marked walkway. Only descriptive analysis done.
Time Frame: Baseline, Month 6 and Month 12
Population: The Full Analysis Set (FAS), which consisted of all participants with an observed value, was considered.
Measure: Mean (Standard Deviation); unit: Meter (m)
Arm/Group | LCZ696 (Sacubitril / Valsartan)
Number analyzed (Participants) | 279
Meter (m)
  Value at Baseline (Day 1) | 392.62 (139.3277)
  Change from Baseline at Month 6: number analyzed (Participants) | 222
  Change from Baseline at Month 6 | 11.99 (67.5725)
  Change from Baseline at Month 12: number analyzed (Participants) | 219
  Change from Baseline at Month 12 | 8.19 (71.3619)

6. Secondary Outcome: Time to Each Up-titration to LCZ696 100 mg and LCZ696 200 mg
Description: To describe the time of up-titration for each dose (24 mg sacubitril / 26 mg valsartan bid and 49 mg sacubitril / 51 mg valsartan bid) of LCZ696. Only descriptive analysis done.
Time Frame: Baseline, Week 2, Week 4, Month 3, Month 6 and Month 12
Population: The Full Analysis Set (FAS), which consisted of all participants with an observed value, was considered.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | LCZ696 (Sacubitril / Valsartan)
Number analyzed (Participants) | 302
Days
  50- 100 mg bid level: number analyzed (Participants) | 248
  50- 100 mg bid level | 21.44 (23.1799)
  100- 200 mg bid level: number analyzed (Participants) | 224
  100- 200 mg bid level | 27.37 (28.5601)
  50- 200 mg bid level: number analyzed (Participants) | 200
  50- 200 mg bid level | 46.61 (36.9439)

7. Secondary Outcome: Median Time to Reach LCZ696 200 mg
Description: as for outcome 6
Time Frame: Baseline, Week 2, Week 4, Month 3, Month 6 and Month 12
Population: The Full Analysis Set (FAS), which consisted of all participants with an observed value, was considered.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | LCZ696 (Sacubitril / Valsartan)
Number analyzed (Participants) | 302
Days | 37.00 [35.00 to 42.00]

8. Secondary Outcome: Percentage of Participants on Guideline Recommended Dose of Beta-blockers and MRAs Over Time
Description: To describe the adherence to guideline recommended dosing of beta-blockers and MRAs at 6 and 12 months of treatment of LCZ696. Only descriptive analysis done.
Time Frame: Baseline, Month 6 and Month 12
Population: The Safety Analysis Set (FAS), which consisted of all participants with an observed value, was considered.
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 (Sacubitril / Valsartan)
Number analyzed (Participants) | 302
Participants
  Baseline | 298
  Month 6 | 272
  Month 12 | 261

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately 1 year.
Arm/Group | LCZ696 (Sacubitril / Valsartan)
All-Cause Mortality (participants affected / at risk) | 9/302
Serious Adverse Events (participants affected / at risk) | 47/302
Other Adverse Events (participants affected / at risk) | 98/302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 (Sacubitril / Valsartan) (N=302)
Anaemia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 3
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Atrial tachycardia (Cardiac disorders) | 1
Bradyarrhythmia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 3
Cardiac failure (Cardiac disorders) | 3
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 13
Congestive cardiomyopathy (Cardiac disorders) | 1
Nodal arrhythmia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Volvulus (Gastrointestinal disorders) | 1
Death (General disorders) | 3
Multiple organ dysfunction syndrome (General disorders) | 1
Sudden death (General disorders) | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1
Bacteraemia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Infective exacerbation of bronchiectasis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Pneumococcal sepsis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 6
Postoperative wound infection (Infections and infestations) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Brain natriuretic peptide increased (Investigations) | 1
White blood cell count increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Fluid overload (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Intracranial mass (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Device malfunction (Product Issues) | 1
Adjustment disorder (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 1
Laryngeal mass (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 (Sacubitril / Valsartan) (N=302)
Diarrhoea (Gastrointestinal disorders) | 18
Fatigue (General disorders) | 19
Dizziness (Nervous system disorders) | 45
Cough (Respiratory, thoracic and mediastinal disorders) | 20
Hypotension (Vascular disorders) | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-07-04): https://cdn.clinicaltrials.gov/large-docs/74/NCT02690974/SAP_000.pdf
  • Study Protocol (2016-09-12): https://cdn.clinicaltrials.gov/large-docs/74/NCT02690974/Prot_001.pdf